CLINICAL TRIAL: NCT03258125
Title: Expression of miRNA-452 in Patients With Early Onset Preeclampsia and Its Correlation With MMP-9
Brief Title: miRNA-452 in Patients With Preeclampsia and Its Correlation With MMP-9
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, FYAli, principal investigator, Assiut University
Other Study IDs: miR-452PE
Record Dates: First submitted 2017-08-20; First posted 2017-08-23 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Real-Time Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- severe EOPE: EOPE: PE starting before 34 weeks gestation Severe PE (Blood pressure more than 160/ 110 mm Hg on 2 occasions 2 hours to 2 weeks apart and proteinuria ( 24-hour urine protein >2000 mg/d).
  Interventions: Genetic: real time PCR (rPCR)
- control: Healthy Pregnant women who come for termination of pregnancy by vaginal delivery or CS between 28-34 weeks gestational age.
  Interventions: Genetic: real time PCR (rPCR)

INTERVENTIONS:
Genetic: real time PCR (rPCR) — A villus tissue (2.5 cm * 2.5 cm * 2.5 cm) will be cut off immediately from the center of placenta, avoiding the area of infarction, bleeding or calcification. After being washed with normal saline, the tissue will be preserved in liquid nitro¬gen at once for subsequent detection of miR-452 and MMP-9 expression by real time PCR (r-PCR). During this procedure total RNA will be extracted including miR-452 and mRNA of MMP-9. Then by reverse transcriptase RNA will be converted into DNA which will be amplification during the PCR, i.e. in real-time, and not at its end, as in conventional PCR. Expression of miR-452 and MMP-9 will be estimated and correlated with each other.

SUMMARY:
Preeclampsia is a pregnancy related disease characterized by the new onset of hypertension and proteinuria after 20 weeks of gestation in previously normotensive women. PE is one of the most challenging diseases in obstetrics worldwide that affects 2-8 % of pregnancies causing both morbidity and mortality of both mother and fetus.

DETAILED DESCRIPTION:
The etiology and pathophysiology of preeclampsia are still unclear but the impaired invasive ability of the trophoblast cells of the placenta and vascular endothelial cell damage are the main two factors. The invasiveness of trophoblast cells depends on the production of proteases, particularly matrix metalloproteinases (MMP). MMPs are a family of 24 zinc dependent endopeptidases capable of degrading extra cellular matrix components. MMP-9 plays an important role in placental invasion and implantation.

MicroRNAs (miRs) are a class of small (19-24 nucleotides in length), single-stranded, non-protein-coding RNAs, which suppress translation or promote the degradation of target messenger RNAs (mRNAs) and thus play an important role in the regulation of cell proliferation, differentiation, apoptosis and even development of cancer.

The role of miRNA in preeclampsia pathogenesis has been investigated in a number of studies. One of the target areas of the miRNAs that forms a link with preeclampsia pathogenesis is the dysregulation of trophoblast differentiation, proliferation, and invasion; this occurs during early pregnancy and leads to the development of preeclampsia; a range of miRNAs have been confirmed to play pivotal roles in these processes by targeting a number of different genes.

MiR-452 is a newly discovered cancer related type of miRNA that was shown to be involved in invasion process where it was upregulated in certain types of cancer such as blad¬der cancer, urothelial carcinoma, and hepatocellular carcinoma and was found to be significantly decreased in other types of cancer such as non-small cell lung cancer , glioma, prostate cancer and Gastric cell cancer.

Based on these previous studies which demonstrate the effect of miR-452 in invasion process of cancer cells either by stimulation or inhibition and that preeclampsia is a disease of impaired placental invasion in which MMP-9 play an important role, we will investigate the placental tissues expression changes of miR-452 which is not studied yet in early onset preeclampsia patients compared to control and try to find a possible mechanism by which it act on placental invasion by measuring expression level of MMP-9 and making correlation between them. The results of this study will provide experimental and theo¬retical basis for clinical prediction, prevention and treatment of preeclampsia.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who come for termination of pregnancy by vaginal delivery or CS between 28-34 weaks gestational age in Assiut university maternity hospital in the age range of 18-40 years.

Exclusion Criteria:

* 1) Diabetes mellitus 2) Chronic hypertension 3) Nephropathy 4) Acute or chronic infectious diseases or other chronic illness 5) Twins pregnancy 6) Anti phospholipid antibody syndrome 7) PE complicated with eclampsia, DIC or HELP syndrome

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women coming for delivery.
Study Population: Pregnant women who come for termination of pregnancy by vaginal delivery or CS between 28-34 weaks gestational age in Assiut university maternity hospital in the age range of 18-40 years.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Expression of miRNA-452 and MMP-9. | one year
  real time polymerase chain reaction

SECONDARY OUTCOMES:
Differences in placental and neonatal weight between the two groups | one year
  weight the placenta and fetus in kilograms

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abbas, MD, Study Director — Assiut University
Locations (1):
- Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No